CLINICAL TRIAL: NCT02074124
Title: Abdominal Tissue Perfusion Changes in Esophageal and Gastric Cancer During Adenosine Vasodilation Measured With Computed Tomography (CT) Perfusion
Brief Title: CT Perfusion Changes in GI Cancer During Adenosine Vasodilation Test
Status: Completed | Type: Observational
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Martin Lundsgaard Hansen, MD, Rigshospitalet, Denmark
Other Study IDs: H-3-2012-067; H-3-2012-067 (Other: Committees on Biomedical Research for the Capital Region of Denmark)
Record Dates: First submitted 2014-02-20; First posted 2014-02-28 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Esophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adenosine Vasodilation test: Group scanned with CT perfusion during adenosine vasodilation test.
- Reference group: Group scanned twice without adenosine vasodilation test for a reference. No randomization.

SUMMARY:
The aim of this study was to investigate changes in abdominal tissue perfusion during adenosine vasodilation. Our hypotheses were that CT perfusion measurements are altered by changes in the circulatory system mediated by adenosine, and a more differentiated assessment of the circulatory capacity of abdominal tumours could be achieved by sequential rest and adenosine vasodilation CT perfusion measurements.

ELIGIBILITY:
Inclusion Criteria:

* Tumour larger than 1.5 cm on diagnostic CT
* Normal serum creatinine
* Age above 18
* Informed written and oral consent.

Exclusion Criteria:

* Contrast allergy or contrast induced nephropathy
* BMI > 40
* Asthma or Chronic Obstructive Lung Disease
* Heart failure (NYHA III+)
* Heart conduction disorder
* Atrial fibrillation
* 2nd/3rd Heart block
* Long QT syndrome
* Wolf Parkinson White Syndrome
* Moderate / severe aortic stenosis
* Haemodynamic contraindications for adenosine, systolic pressure below 90

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven tumors in esophagus or stomach
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in arterial flow during adenosine vasodilation test (CT perfusion parameter) | 0 min and 15 min

SECONDARY OUTCOMES:
Change in Blood pressure during adenosine vasodilation test | 0 min and 15 min
Change in Heart rate during adenosine vasodilation test | 0 min and 15 min
Change in Area under arterial input curve during adenosine vasodilation test | 0 min and 15 min
  Area Under Curve (AUC) is correlated to cardiac output
Change in Blood volume (CT perfusion parameter) during adenosine vasodilation test | 0 min and 15 min
Change in Permeability (CT perfusion parameter) during adenosine vasodilation test. | 0 min and 15 min

CONTACTS AND LOCATIONS:
Overall Officials: Martin L Hansen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark